CLINICAL TRIAL: NCT02126969
Title: A Phase II Study of Docetaxel, Carboplatin With and Without Low Dose Radiation as Induction Therapy in Locally Advanced Head and Neck Cancer
Brief Title: A Study of Chemo +/- Low-dose Radiation as Induction Therapy in SCCHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susanne Arnold (Other)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCC-13-HN-24
Record Dates: First submitted 2014-04-23; First posted 2014-04-30 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer; Larynx
Keywords: Cancer; Low dose radiation
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases; Neoplasms | interventions — Drug Therapy; Docetaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy plus Radiation Therapy (Experimental): Low dose fractionated radiation - 80cGy with chemotherapy
  Interventions: Radiation: Low dose fractionated radiation - 80cGy with chemotherapy
- Chemotherapy without Radiation (Active Comparator): Chemotherapy only
  Interventions: Drug: Docetaxel and Carboplatin AUC 6

INTERVENTIONS:
Radiation: Low dose fractionated radiation - 80cGy with chemotherapy — Chemotherapy + 80 cGy of RT
  Arms: Chemotherapy plus Radiation Therapy
Drug: Docetaxel and Carboplatin AUC 6 — Docetaxel 75 mg/m2 and Carboplatin AUC 6 without Radiation
  Arms: Chemotherapy without Radiation

SUMMARY:
The primary hypothesis of this study is that hyper-radiosensitivity (HRS) seen at extremely low doses of radiation can be exploited to enhance the effect of chemotherapy, and that this effect differs from the cellular effect of higher, standard fractions of radiation used in traditional radiation treatment paradigms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced head and neck cancer of squamous type stage III, IVA and IV B and select Stage II tumors of the BOT who are appropriate for potentially curative therapy with chemoradiotherapy.
* Measurable disease.
* ECOG performance status of 0, 1 or 2
* No prior chemotherapy for the current locally advanced SCCHN.
* Age ≥18 years.
* Life expectancy of greater than 3 months
* Normal organ and marrow function measured within 14 days of registration as defined below:

  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin < institutional upper limit of normal
  * AST(SGOT ≤ 2.5 × institutional upper limit of normal
  * Alkaline phosphatase ≤ 2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits
* OR

  o Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, throughout the duration of active treatment and for 4 months after completion of chemotherapy and radiation. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of active study treatment, and for 4 months after completion of chemotherapy and radiation (both induction and definitive) administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior chemotherapy for SCCHN
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Carboplatin or Docetaxel.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women
* HIV-positive patients on combination antiretroviral therapy
* Other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated previous Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 3 years.
* Patients with nasopharynx or salivary gland primary site
* Patients with distant metastatic disease (M1c)
* Patients with grade II or greater peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Arnold, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy Plus Radiation Therapy | Chemotherapy Without Radiation
Started | 23 | 22
Completed | 22 | 20
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Plus Radiation Therapy | Chemotherapy Without Radiation | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (6.7) | 55 (8.1) | 57 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 21 | 44
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Primary Site Complete Response Rate
Description: Primary site is defined as the original, or first site that the cancer developed in the body. In this study, primary sites within the head and neck included squamous cancers of the larynx, oral cavity, oropharynx, hypopharynx.Complete response rate in patients treated with 2 cycles of induction Docetaxel and Carboplatin with low dose fractionated radiation therapy (LDFRT) will be compared to those treated with chemotherapy alone. CRR was determined Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Where possible, surgeon also evaluated primary site and provided response assessment.
Time Frame: Up to 50 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Radiation Therapy | Chemotherapy Without Radiation
Number analyzed (Participants) | 22 | 20
Participants | 6 | 4

2. Secondary Outcome: Overall Response Rate
Description: To assess overall response rate of patients to 2 cycles of induction Docetaxel and Carboplatin with or without LDFRT. Response assessment was Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, and Progressive Disease (PD): > 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 50 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Radiation Therapy | Chemotherapy Without Radiation
Number analyzed (Participants) | 22 | 20
Participants
  Overall Complete Response Rate | 1 | 1
  Overall Partial Response Rate | 11 | 12
  Overall Stable Disease Rate | 10 | 7
  overall Progressive Disease Rate | 0 | 0

3. Secondary Outcome: Change in Quality of Life (QOL) of Patients Receiving Low Dose Fractionated Radiation Therapy With Chemotherapy.
Description: Quality of Life (QOL) will be measured pre- and post-treatment using a single 5-question QOL well-being survey. The change in score will be presented independently for each subpart of the QOL survey.
  1. Physical; scores range from 7-35; higher scores indicate increased well-being
  2. Social/family; scores range from 7-35; higher scores indicate increased well-being
  3. Emotional; scores range from 6-30; higher scores indicate increased well-being
  4. Functional; scores range from 7-35; higher scores indicate increased well-being
  5. Additional Concerns; scores range from 10-50; lower scores indicate increased well-being
  6. FACT-G is the sum of the first 4 scores; scores range from 27-135; higher scores indicated increased well-being
  7. FACT-H&N is the sum of the first five scores; scores range from 37-185; higher scores indicated increased well-being
  8. Trial Outcome Index is the sum of 1, 4 and 5; scores range from 24-120; higher scores indicated increased well-being
Time Frame: Up to 50 days (pre- and post-treatment)
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | Chemotherapy Plus Radiation Therapy | Chemotherapy Without Radiation
Number analyzed (Participants) | 22 | 20
change in score
  PHYSICAL WELL-BEING SCORE | -1.46 (5.12) | -1.64 (7.22)
  SOCIAL/FAMILY WELL-BEING SCORE | -1.34 (4.55) | -2.34 (3.72)
  EMOTIONAL WELL-BEING SCORE | 2.05 (3.75) | 1.60 (4.31)
  FUNCTIONAL WELL-BEING SCORE | -0.48 (6.04) | -1.70 (4.92)
  FACT-G TOTAL SCORE | -1.23 (13.52) | -4.08 (12.72)
  ADDITIONAL CONCERNS SCORE | 5.01 (8.24) | 3.63 (7.80)
  FACT-H&N TOTAL SCORE | 3.79 (18.05) | -0.46 (19.16)
  TRIAL OUTCOME INDEX SCORE | 3.08 (14.55) | 0.29 (15.05)

4. Secondary Outcome: 3-year Overall Survival
Description: 3-year overall survival
Time Frame: From date of randomization until date of death from any cause, assessed up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Radiation Therapy | Chemotherapy Without Radiation
Number analyzed (Participants) | 22 | 20
Participants | 14 | 11

ADVERSE EVENTS:
Time Frame: The first subject on was randomized on 1/30/2015 and last subject was randomized on 2/26/2018. Data was collected for AE reporting during treatment and following treatment to the first interval scans, thus AE collection occurred over approximately a 6 month period from randomization to the end of treatment for each subject, mortality assessed up to 3 years.
Arm/Group | Chemotherapy Plus Radiation Therapy | Chemotherapy Without Radiation
All-Cause Mortality (participants affected / at risk) | 8/22 | 9/20
Serious Adverse Events (participants affected / at risk) | 12/22 | 6/20
Other Adverse Events (participants affected / at risk) | 22/22 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Plus Radiation Therapy (N=22) | Chemotherapy Without Radiation (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 5 (6) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 1 (1)
White blood cell decreased (Investigations) | 4 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Plus Radiation Therapy (N=22) | Chemotherapy Without Radiation (N=20)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 7 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 5 (6) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 5 (6) | 6 (6)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 11 (11) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 4 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 5 (6)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 18 (53) | 18 (41)
Nausea (Gastrointestinal disorders) | 16 (24) | 16 (24)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (19) | 9 (11)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (10) | 9 (11)
Fever (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 3 (3) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 10 (12) | 6 (8)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 14 (20) | 12 (19)
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (6) | 3 (6)
Neutrophil count decreased (Investigations) | 11 (15) | 4 (5)
Platelet count decreased (Investigations) | 2 (2) | 1 (3)
Weight loss (Investigations) | 1 (3) | 5 (6)
White blood cell decreased (Investigations) | 9 (12) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (3)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (5)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT02126969/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT02126969/ICF_001.pdf